CLINICAL TRIAL: NCT06812260
Title: A Single-arm, Open-label, Phase II Study to Evaluate Clinical Efficacy, Safety and Pharmacokinetics of HLX10 (Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection) in Combination With Chemotherapy (Carboplatin-Etoposide) in Previously Untreated Japanese Patients With Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: A Single-arm, Open-label, Phase II Study to Evaluate Efficacy, Safety and Pharmacokinetics of HLX10 + Chemotherapy in Patients With ES-SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10-005-SCLC301JP; entered later (Other: jRCT)
Record Dates: First submitted 2025-01-22; First posted 2025-02-06 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: SCLC, Extensive Stage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): HLX10 + Chemotherapy (Carboplatin- Etoposide)
  Interventions: Drug: HLX10+chemo

INTERVENTIONS:
Drug: HLX10+chemo — Treatment arm

SUMMARY:
Evaluate Clinical Efficacy, Safety and Pharmacokinetics of HLX10 (Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection) in Combination with Chemotherapy (Carboplatin-Etoposide) in Previously Untreated Japanese Patients with Extensive Stage Small Cell Lung Cancer (ES-SCLC)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in clinical studies; fully understand, be informed about the study and have signed the informed consent form (ICF); willingness to follow and ability to complete all trial procedures.
2. Male or female aged ≥ 18 years at the time of signing the ICF.
3. Histologically or cytologically diagnosed with ES-SCLC (according to the Veterans Administration Lung Study Group staging system).
4. No prior systemic therapy for ES-SCLC (including systemic chemotherapy, molecular targeted therapy, biological therapy, and other investigational therapies, etc.).
5. Subjects who have received chemoradiotherapy for previous limited stage SCLC must be treated with curative intent and have a treatment-free interval of at least 6 months from the last course of chemotherapy, radiotherapy, or chemoradiotherapy to the diagnosis of extensive stage SCLC.
6. At least one measurable lesion as assessed by the IRRC according to RECIST 1.1 within 4 weeks prior to first dose.

Exclusion Criteria:

1. Histologically or cytologically confirmed mixed SCLC.
2. Other active malignancies within 5 years or at the same time. Localized tumors that have been cured, such as basal cell carcinoma, squamous-cell skin cancer, superficial bladder cancer, prostate carcinoma in situ, cervical cancer in situ and breast cancer in situ are acceptable.
3. Subjects who are preparing for or have received an organ or bone marrow transplant.
4. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Subjects with indwelling catheters are allowed regardless of drainage frequency.
5. Subjects with known or documented active CNS metastases and/or carcinomatous meningitis at screening. However, the following subjects are allowed to be enrolled: 1) Subjects with asymptomatic brain metastases (i.e., no progressive central nervous system symptoms caused by brain metastases, no requirement for corticosteroids, and lesion size ≤ 1.5 cm) may be included, but are required to receive regular brain imaging as a site of lesion. 2) Subjects with treated brain metastases which have been stable for at least 2 months (as confirmed by 2 radiological examinations at least 4 weeks apart after treatment of brain metastases), with no evidence of new or enlarging brain metastases, and with discontinued steroids 3 days prior to study drug administration. (Stable brain metastases here should be confirmed before the first dose of the study drug.).
6. Subjects with spinal cord compression that has not been radically treated with surgery and/or radiotherapy.
7. Subjects with myocardial infarction within half a year before the first dose of the study drug, poorly controlled arrhythmia (including QTc intervals ≥ 450 ms for males and ≥ 470 ms for females) (QTc intervals are calculated by Fridericia's formula).
8. Class III to IV cardiac insufficiency according to NYHA classification or a left ventricular ejection fraction < 50% by cardiac color Doppler.
9. Subject has uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN).
10. Subject with peripheral neuropathy ≥ Grade 2 by CTCAE.
11. Human immunodeficiency virus (HIV) infection, positive test for HIV antibody.
12. Active or latent pulmonary tuberculosis.
13. Subjects with previous and concurrent interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis and severe impaired pulmonary function that may interfere with the detection and management of suspected drug-related pulmonary toxicity, as judged by the investigator.
14. Hepatitis B (positive test for HBsAg or HBcAb and positive test for HBV-DNA) or Hepatitis C (positive tests for HCV antibody and HCV-RNA). Hepatitis B and C coinfection (positive test for HBsAg or HBcAb and positive test for HCV antibody).
15. Known active or suspected autoimmune diseases. Subjects in a stable state with no need for systemic immunosuppressant therapy are allowed to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Response (CR or PR) rate at week 24 | up to 2 years
  Response (CR or PR) rate at week 24 (assessed by independent radiology review committee [IRRC] based on Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)

SECONDARY OUTCOMES:
Overall survival (OS) | up to 3 years
PFS (assessed by the IRRC and investigator based on RECIST 1.1) | up to 3 years
Objective response rate (ORR) (assessed by the IRRC and investigator based on RECIST 1.1) | up to 3 years
Duration of response (DOR) (assessed by the IRRC and investigator based on RECIST 1.1) | up to 3 years
safety | up to 3 years
  Adverse events (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Kansai Medical University Hospital Department of Respiratory Oncology, Hirakata, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No